CLINICAL TRIAL: NCT00931450
Title: Pilot / Phase II Randomised, Double Blind, Placebo Controlled Multicenter Study With Biomarker Evaluation of Neoadjuvant Exemestane in Combination With Sunitinib in Post-menopausal Women With Hormone- Sensitive, Her-2 Negative Primary Breast Cancer.
Brief Title: Sunitinib Malate and Exemestane in Treating Postmenopausal Women With Breast Cancer
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Institut Català d'Oncologia (Other)
Organization: National Cancer Institute (NCI) (NIH)
Allocation: Randomized | Masking: Double | Purpose: Treatment
Other Study IDs: ICO-SUT-EXE-08; CDR0000640330 (Registry Identifier: PDQ (Physician Data Query)); PFIZER-ICO-SUT-EXE-08
Record Dates: First submitted 2009-07-01; First posted 2009-07-02 (Estimated); Last update posted 2013-08-12 (Estimated); Status verified 2009-07

CONDITIONS: Breast Cancer
Keywords: estrogen receptor-positive breast cancer; HER2-negative breast cancer; stage IA breast cancer; stage IB breast cancer; stage II breast cancer; stage IIIA breast cancer; stage IIIB breast cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — exemestane; Sunitinib

ARMS (2):
- Group 1 (Active Comparator): Patients receive oral exemestane and oral placebo once daily on days 1-28. Treatment repeats every 4 weeks for 6 courses in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: exemestane; Other: placebo
- Group 2 (Experimental): Patients receive oral exemestane once daily and oral sunitinib malate once daily on days 1-28. Treatment repeats every 4 weeks for 6 courses in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: exemestane; Drug: sunitinib malate

INTERVENTIONS:
Drug: exemestane — Given orally
Drug: sunitinib malate — Given orally
  Arms: Group 2
Other: placebo — Given orally
  Arms: Group 1

SUMMARY:
RATIONALE: Sunitinib malate and exemestane may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth. Giving sunitinib malate and exemestane before surgery may make the tumor smaller and reduce the amount of normal tissue that needs to be removed.

PURPOSE: This randomized phase I/II trial is studying the side effects and best dose of sunitinib malate to see how well it works when given together with exemestane in treating postmenopausal women with breast cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Determine the safe dose level of sunitinib malate that can be combined with exemestane (pilot phase I).
* Evaluate the clinical response of neoadjuvant therapy comprising exemestane and sunitinib malate in postmenopausal women with hormone receptor-positive and HER-2 negative primary breast cancer (phase II).

Secondary

* Evaluate the safety and feasibility of this regimen in these patients.
* Evaluate the percentage of patients undergoing breast-conserving surgery after completion of study therapy.
* Determine the safety profile of this regimen in these patients.
* Determine the rate of complete pathological response in the breast and axillary lymph nodes at the time of surgery.
* Determine the extent of treatment-related inhibition of phosphorylation of VEGFR-2, PDGF, and c-KIT receptor tyrosine kinases.
* Find a genetic profile, based on the analysis of CYP19A1 polymorphisms, able to predict response to exemestane in neoadjuvant setting.
* Conduct exploratory investigation of biomarkers expression before and during therapy in order to identify molecular characteristics of responding tumors.

OUTLINE: This is a multicenter, dose-escalation study of sunitinib malate followed by a phase II study.

* Phase I pilot: Patients receive oral sunitinib malate and oral exemestane once daily on days 1-28. Treatment repeats every 4 weeks for 6 courses in the absence of disease progression or unacceptable toxicity.
* Phase II: Patients are randomized to 1 of 2 treatment groups:

  * Group 1: Patients receive oral exemestane and oral placebo once daily on days 1-28. Treatment repeats every 4 weeks for 6 courses in the absence of disease progression or unacceptable toxicity.
  * Group 2: Patients receive oral exemestane once daily and oral sunitinib malate once daily on days 1-28. Treatment repeats every 4 weeks for 6 courses in the absence of disease progression or unacceptable toxicity.

At 7-15 days after completion of study therapy, patients undergo definitive surgery.

Blood and tissue samples are collected at baseline and periodically during study to examine inhibition of phosphorylation of VEGFR-2, PDGF, and c-KIT receptor tyrosine kinases; CYP19A1 polymorphisms; and biomarkers analysis by cDNA microarrays, ELISA, and RT-PCR.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed invasive breast carcinoma meeting the following criteria:

  * Estrogen receptor-positive ≥ 50% or Allred score > 6
  * HER-2 negative defined as IHC < 2+ and negative FISH/CISH
  * Primary tumor measuring ≥ 3 cm if there is no node involvement
  * Any T if N1 or N2 disease

    * No inflammatory breast cancer (T4d)
  * No metastatic disease
* Measurable disease by mammography and/or ultrasound and MRI (if available)

PATIENT CHARACTERISTICS:

* Postmenopausal

  * Prior bilateral oophorectomy
  * ≥ 60 years of age
  * < 60 years of age AND have experienced amenorrhea for ≥ 12 months in the absence of chemotherapy, tamoxifen, or toremifene OR have undergone ovarian suppression and follicle-stimulating hormone and estradiol levels in the postmenopausal range
* ECOG performance status 0-1
* ANC ≥ 1,500/mm^3
* Platelet count ≥ 100,000/mm^3
* Hemoglobin ≥ 10 g/dL
* Serum creatinine ≤ 1.5 mg/dL OR creatinine clearance ≥ 50 mL/min
* Bilirubin normal
* AST and ALT ≤ 2.5 times upper limit of normal (ULN)
* Alkaline phosphatase ≤ 2.5 times ULN
* Albumin > 2.5. g/dL
* No known HIV infection
* Adequate left ventricular ejection fraction (LVEF) at baseline defined as LVEF not below normal range by echocardiogram or MUGA
* No evidence of prior uncontrolled hypertension

  * Patients with controlled hypertension (systolic < 150 mm Hg and/or diastolic < 90 mm Hg) by antihypertensive therapies allowed
* No prior uncontrolled or symptomatic angina, myocardial infarction, congestive heart failure, clinically significant arrhythmias, or prolongation of the QTc interval
* No hemorrhagic or thrombotic events, including transient ischemic attack, pulmonary embolism, or deep-vein thrombosis, within the past 12 months
* No gross hemorrhage within the past 6 months (e.g., gastrointestinal bleeding, hemoptysis, or hematuria)
* No history or evidence of an inherited bleeding diathesis or coagulopathy at risk of bleeding
* None of the following:

  * Unable to swallow oral medications
  * Active inflammatory bowel disease
  * Partial or complete bowel obstruction
  * Chronic diarrhea
* No history of another malignancy within the past 5 years except for cured non-melanoma skin cancer or successfully treated carcinoma in situ of the cervix
* No psychiatric disease or social situations that would limit compliance with study requirements or patient unwilling or unable to comply with protocol for the duration of study
* No unstable or severe intercurrent medical condition that, in the opinion of the investigator, might interfere with the achievement of study objectives
* No known immediate or delayed hypersensitive reaction or idiosyncrasy to drugs chemically related to exemestane or sunitinib malate or their excipients

PRIOR CONCURRENT THERAPY:

* See Disease Characteristics
* No prior or other concurrent chemotherapy, radiotherapy, immunotherapy, biologic therapy, or hormonal therapy for primary invasive breast cancer
* No concurrent anticoagulant therapy except for low-dose anticoagulants (i.e., low molecular weight heparin or aspirin) for the prevention of deep-vein thrombosis
* No chronic therapy with corticosteroids, except for steroids administered by inhalation
* More than 4 weeks since prior major surgery and ≥ 7 days since prior minor surgery
* No prior or other concurrent investigational anticancer agent
* No concurrent participation in another clinical trial
* No concurrent drugs with potential proarrhythmic activity
* No concurrent known CYP3A4 inhibitors (i.e., grapefruit, verapamil, ketoconazole, miconazole, itraconazole, erythromycin, clarithromycin, diltiazem, nefazodone, voriconazole, telithromycin, indinavir, saquinavir, ritonavir, nelfinavir, delavirdine)
* No concurrent known CYP3A4 or CYP1A2 inducers (i.e., carbamazepine, dexamethasone, felbamate, omeprazole, efavirenz, tipranavir, phenobarbital, phenytoin, primidone, rifabutin, rifampicin, St. John's wort)

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2009-03; Primary Completion 2011-10 (Estimated)

PRIMARY OUTCOMES:
Recommended dose of sunitinib malate that can be combined with exemestane
Objective clinical response (complete or partial response) according to WHO criteria

SECONDARY OUTCOMES:
Safety and feasibility of the combination of sunitinib malate and exemestane
Safety profile
Rate of breast-conserving surgery
Percentage of pathological complete response in the breast and axillary lymph nodes
Grade of inhibition of phosphorylation of VEGFR-2, PDGF, and c-KIT receptor tyrosine kinases
Genetic profile, based on the analysis of CYP19A1 polymorphisms, able to predict response to neoadjuvant exemestane
Molecular biomarkers predictive of response

CONTACTS AND LOCATIONS:
Overall Officials: Sonia Pernas, MD — Institut Català d'Oncologia
Locations (1):
- Institut Catala D'Oncologia, L'Hospitalet de Llobregat, Spain

REFERENCES:
- [Derived] Fullana B, Morales S, Petit A, Alay A, Verdaguer H, Climent F, Navarro-Perez V, Cejuela M, Galvan P, Guma A, Llombart-Cussac A, Cordero D, Casanovas O, Prat A, Gil-Gil M, Pernas S. Neoadjuvant sunitinib plus exemestane in post-menopausal women with hormone receptor-positive/HER2-negative early-stage breast cancer (SUT_EXE-08): a phase I/II trial. Sci Rep. 2024 Oct 9;14(1):23626. doi: 10.1038/s41598-024-72152-1. PMID 39384801